CLINICAL TRIAL: NCT01154465
Title: Impact of Ultrasound Guided Central Venous Catheterization on Complications in Obese Patients in Intensive Care Unit
Brief Title: A Trial to Study the Influence of Ultrasound Guidance on the Complications of Central Catheter
Acronym: CATHETER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOL09-PR-DUPONT; 2009-A01335-52 (Other: RCB)
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Central Venous Catheters; Obesity
Keywords: Central venous catheterization; Obese; Ultrasound guidance; Jugular; Randomized; Intensive Care Unit
MeSH Terms: conditions — Obesity | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anatomical guidance puncture (Active Comparator): The patient is placed supine (with a slight neck extension for jugular punctures).
  The preparation of the CVC installation will follow the procedures for disinfection, for skin preparation of the operator, for installation of sterile fields and for local anaesthesia.
  The veins will be tracked by simple palpation of the carotid pulse.
  The puncture will be made following:
  * The anterior Boulanger's incision for the internal jugular vein;
  * When venous aspiration is obtained, the catheter is assembled according to the Seldinger method.
  Interventions: Procedure: Central Venous Catheter Insertion
- US-guided puncture (Experimental): The patient is placed supine (with a slight neck extension for jugular punctures).
  The ultrasound probe will be isolated by a sterile protective plastic and the operator will mount a ramp on which the puncture syringe needle is placed. A sterile gel will be used in order to visualize the vein and directly puncture under ultrasound guidance following:
  - The anterior Boulanger's incision for the internal jugular vein pathway;
  Interventions: Procedure: Central Venous Catheter Insertion; Device: Ultrasound guidance

INTERVENTIONS:
Procedure: Central Venous Catheter Insertion — The preparation of the CVC installation will follow the procedures for skin preparation of the operator, installation of sterile fields and local anaesthesia.
  The patients' skin disinfection before catheter insertion and care will follow the protocol:
  * Clean the area of insertion of the catheter with a solution of 4% aqueous povidone foaming (Betadine Scrub).
  * Rinse with sterile water and then drying.
  * First application of 5% alcohol povidone-iodine (alcoholic Betadine) far beyond the area of insertion.
  * Second application of 5% alcoholic povidone-iodine (alcoholic Betadine) by the operator after sterile draping.
  After sterilisation and puncture, the Seldinger technique is employed to insert the line: a blunt guidewire is passed through the needle, and the needle is then removed.
  Other Names: Betadine; Arrow®
Device: Ultrasound guidance — The ultrasound probe will be isolated by a sterile protective plastic and the operator will mount a ramp on which the puncture syringe needle is placed.
  A sterile gel will be used in order to visualize the vein and directly puncture under ultrasound guidance following:
  - The anterior Boulanger's incision for the internal jugular vein When venous aspiration is obtained, the needle can easily be removed from the ramp and the syringe to mount the catheter following Seldinger's method.
  Other Names: Site~Rite ® V (C.R. Bard Inc)
  Arms: US-guided puncture

SUMMARY:
Central venous catheterization (CVC) in ICU is very common. It is associated with many complications. These complications are now well identified in the literature. They are primarily mechanical, infectious and thrombotic events. Many measures are taken to reduce them as the choice of insertion site, strict aseptic technique during insertion and type of catheter used. However, despite these measures, it appears that the incidence of these complications is still high. The technique of ultra-sound guided (USG) catheter insertion has shown its effectiveness in reducing complications in the general ICU population. The increase in obesity in the general population is accompanied by an increase in the obese population in the ICU (BMI > 30 kg.m-2). Many studies have investigated the effect of obesity on morbidity and mortality in ICU. Some studies found a higher rate of catheter infections in obese patient. Moreover, insertion of central venous catheter is technically more difficult in obese patients.

To the investigators knowledge there are no studies on the impact of USG central venous catheterization in obese patients in ICU.

The objective of this prospective randomized controlled study is to demonstrate the superiority of USG central venous catheterization (jugular or femoral) on complications in a population of obese patients. 450 patients will be included and dispatched in two groups (jugular or femoral) according to the chosen site of catheter insertion. In both groups, patients will be randomized in the USG technique or the usual anatomical technique.

The rate of complications (mechanical, thrombotic or infectious) will be the primary endpoint. Secondary endpoints will be the following: rate of catheter colonization, rate of catheter-related bacteremia, rate of failure during insertion, number of punctures, procedure timing and mortality The investigators hope to establish a benefit in the use of USG central venous catheterization in obese ICU patients and thus contribute to improve the quality of care.

DETAILED DESCRIPTION:
Determination of the insertion technique

The insertion technique (with anatomical landmarks or ultrasound-guided) will be determined by randomization. To that aim, we will use a software available on an intranet server and available from all ICUs involved in the study.

All central venous catheters included in the study will be inserted by experienced physicians trained to the use of ultrasound for the placement of access (minimum 2 previous CVC installations with ultrasound).

The central catheters used in the study (Arrow International, Inc.) are single, double or triple lumen (16 and 20 cm in length). The choice will be made by the clinician in patient management. Catheters impregnated with antibiotics or antiseptics are excluded.

The ultrasound used will be a Site~Rite ® V (C.R. Bard Inc) type equipped with a multifrequency probe of 5-10 MHz.

Acts and examinations performed in the protocol:

* Systematic culture of the CVC and achievement of blood cultures in cases of hyperthermia
* Systematic ultrasound examination at D4 to look for thrombosis.

The examinations and the necessary samples required to the strict follow-up of the patients will be made in the ICUs participating in the study and sent to the usual laboratories for analysis. Ultrasounds will be performed by physicians of the departments participating in the study.

The primary endpoint is the rate of complications related to a composite criterion incorporating mechanical, thrombotic and infectious complications.

The secondary endpoints are:

* Rate of failure / success when placing catheters (failure is defined by three skin biopsies which did not lead to the laying of the venous access).
* The time required for the installation of CVC (time between the first puncture and the introduction of the catheter)
* The number of punctures before final laying
* Type of complications according to the method and site of installation
* The overall mortality according to the technique used
* The duration of stay in ICU / hospital

We define complications as follows:

* Mechanical complications:

  * Number of failed insertion,
  * Number of bleeding which required a compression for more than 30 minutes,
  * Number of arterial wound,
  * Number of misposition visualized on the radiological picture,
  * Rare complications (pneumothorax, hematoma, air embolism).
* Infectious complications (according to the recommendations of the Twelfth Conference of Society Consensus resuscitation French updated in 2002):

  * Colonization of the catheter: Positive culture (≥ 1 000 CFU / ml) according to the quantitative method described by Brun-Buisson of the catheter's distal end (4-5 cm) aseptically removed. This technique can diagnose colonization induced not only by subcutaneous infection, but also by intra vascular pathway. However, it does not differentiate the mode of colonization.
  * Catheter-related infection:

    * In the absence of bacteremia, diagnosis of catheter-related infection will be based on:

      * a positive culture (> 1 000 CFU / ml) and total or partial regression of signs of infection within 48 hours after catheter removal or
      * purulence of the inlet of the catheter or
      * tunnelite.
    * Bacteremic infection related to the C.V.C. will be defined by:

      * the association of one positive bacteremia occurring within 48 hours before or after the withdrawal of CVC (two in case of Staphylococcus epidermidis) and a positive culture of the insertion site by the same organism or a culture of CVC > 1 000 CFU / ml of the same organism or
      * a quantitative central / peripheral blood cultures ratio > 5 or
      * a differential blood culture positivity delay > 2 hours.
    * The infection is NOT related to CVC if :

      * the CVC is finally sterile or
      * the CVC culture is positive, but the strain is different from that isolated in the blood and / or other focus of infection present at the removal of the CVC and sepsis does not regress to the removal of the CVC or
      * the CVC culture is positive and the strain is identical with that found in other infected site found at least 48 hours before removal of the CVC whether or not responsible for bacteremia and sepsis does not regress after the removal of the CVC.
* Thrombotic complications:

A venous Echo-Doppler exploration is performed within four days following the catheter ablation to look for a loss of compressibility of a venous segment under the pressure of the probe associated to an intravascular image measuring more than 3 mm in the anteroposterior diameter (maximum diameter).

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* BMI ≥ 30 kg/m2.
* Patient requiring the installation of a central venous catheter (femoral).
* Informed consent signed.

Exclusion Criteria:

* No particular exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-05-26 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Rate of complications | Within 4 days following installation of CVC
  To compare the rate of complications (mechanical, thrombotic and infectious) of CVC posed by US-guided method vs. anatomical method on obese patients in ICU.

SECONDARY OUTCOMES:
The rate of success/failure installation | Day 1
  Failure rate / success when placing CVC. Failure is defined by three skin biopsies that did not lead to the laying of the venous access.
The time of installation | Day 1
  Time between the first puncture and the correct installation of the catheter
Number of punctures | Day 1
  The number of punctures required to correctly install the CVC
Type of complications | Within 4 days following installation of CVC
  Type of complications depending on the method and site installation
Mortality | Within 4 days following installation of CVC
The duration of stay | Within 4 days following installation of CVC
  The duration of stay in ICU and in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hervé DUPONT, MD-PhD, Principal Investigator — Centre Hospitalo-Universitaire d'Amiens; Norair AIRAPETIAN, MD, Principal Investigator — Centre Hospitalier Universitaire, Amiens
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No